CLINICAL TRIAL: NCT00679848
Title: Transoral Gastric Volume Reduction as an Intervention for Weight Management (TRIM): A Non-Randomized Multicenter Feasibility Study of Subjects With Class II or Low Grade Class III Obesity
Brief Title: Transoral Gastric Volume Reduction as an Intervention for Weight Management
Acronym: TRIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVL-EC-003
Record Dates: First submitted 2008-05-13; First posted 2008-05-19 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Obesity
Keywords: Weight Loss; Transoral Suturing; Experimental
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Transoral Suturing
  Interventions: Device: RS2 (RESTORe Suturing System)

INTERVENTIONS:
Device: RS2 (RESTORe Suturing System) — Suturing in stomach

SUMMARY:
The purpose of this study is to evaluate the safety, technical feasibility, and initial effectiveness (i.e., weight loss primarily measured as percent excess weight loss) of TGVR performed using the Bard RESTORe Suturing System

ELIGIBILITY:
Inclusion Criteria:

* Male, Female; ages >18yrs - £ 60 yrs
* BMI 30-45 kg/m2
* History of obesity for 5 yrs; attempts at weight control ineffective
* Weight stable
* Willing to comply with study requirements
* Agrees to not have any additional weight loss surgery, reconstructive surgery or liposuction for one year following procedure
* Sign informed consent form

Exclusion Criteria:

* Women of childbearing age not practicing effective birth control method or pregnant or lactating
* Mallampati score = 4
* Uncontrolled hypothyroidism
* Previous interventional/surgical treatment of obesity; any prior gastric surgery
* History of diabetes for > 10 yrs or difficult to control diabetes
* Presence of hiatal hernia
* Congenital or acquired anomalies of the GI tract
* Severe cardiovascular, cerebrovascular, or cardiopulmonary disease
* Chronic or acute upper gastrointestinal bleeding conditions
* Helicobacter pylori positive
* Immunocompromised
* Subjects with eating disorders
* Acute or chronic infection
* Significant movement limitations
* Not a candidate for conscious or general anesthesia
* Active substance abuse
* Life expectancy < 2 years
* Enrolled in another investigational drug or device trial that has not completed the primary endpoint or that clinically interferes with this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 24 Months

SECONDARY OUTCOMES:
Technical success of test procedure. | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio